CLINICAL TRIAL: NCT04348812
Title: Transcranial Direct Current Stimulation (tDCS) Augments the Effects of Gamified, Mobile Attention Bias Modification
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: The City College of New York (Other)
Responsible Party: Principal Investigator, Tracy Dennis, Primary Investigator, Hunter College of City University of New York
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 334490
Record Dates: First submitted 2020-04-12; First posted 2020-04-16 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Anxiety; Stress
Keywords: Anxiety, stress
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: All participants received active behavioral intervention combined with either active brain stimulation or sham stimulation control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS Active (Experimental): Transcranial direct current stimulation with ABMT
  Interventions: Behavioral: ABMT; Other: Transcranial direct current stimulation
- tDCS sham (Sham Comparator): Transcranial direct current sham stimulation with ABMT
  Interventions: Behavioral: ABMT

INTERVENTIONS:
Behavioral: ABMT — mobile attention bias modification training for anxiety, using the app Personal Zen
  Other Names: Personal Zen
Other: Transcranial direct current stimulation — Soterix 1X1 tDCS Limited Total Energy (LTE) Stimulator
  Other Names: tDCS
  Arms: tDCS Active

SUMMARY:
The present study tested whether transcranial direct current stimulation (tDCS) across the prefrontal cortex (PFC), versus sham stimulation, effectively augments the beneficial effects of a gamified attention bias modification training (ABMT) mobile app.

DETAILED DESCRIPTION:
Anxiety-related attentional bias (AB) is the preferential processing of threat observed in clinical and sub-clinical anxiety. Attention bias modification training (ABMT) is a computerized cognitive training technique designed to systematically direct attention away from threat and ameliorate AB, but mixed and null findings have highlighted gaps in our understanding of mechanisms underlying ABMT and how to design the most effective delivery systems. One neuromodulation technique, transcranial direct current stimulation (tDCS) across the prefrontal cortex (PFC) may augment the effects of ABMT by strengthening top-down cognitive control processes, but the evidence base is limited and has not been generalized to current approaches in digital therapeutics, such as mobile applications. The present study tested whether tDCS across the PFC, versus sham stimulation, effectively augments the beneficial effects of a gamified ABMT mobile app. Thirty-eight adults (Mage = 23.92, SD = 4.75; 18 females) evidencing low-to-moderate anxiety symptoms were randomly assigned to active or sham tDCS for 30-minutes while receiving ABMT via a mobile app. Participants reported on potential moderators of ABMT, including life stress and trait anxiety. ECG was recorded during a subsequent stressor to generate respiratory sinus arrhythmia (RSA) suppression as a metric of stress resilience.

ELIGIBILITY:
Inclusion Criteria:

* mild - moderate anxiety

Exclusion Criteria:

* psychotic disorder
* substance use disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Self-reported negative mood symptoms | Day 1
  Self report using the Depression, Anxiety, Stress Scale (DASS); Higher scores mean more severe negative mood/worse outcomes (scores ranging from 0-42)
Self-reported subjective state anxiety | Day 1
  Self report of state anxiety using the State-Trait Anxiety Inventory (STAI); Higher scores mean greater anxiety severity/worse outcomes (scores ranging from 20-80).
Threat bias, or dsyregulated attention towards threat, measured via computer assay | Day 1
  Using the computerized, reaction time-based cognitive assessment task, the "dot probe", biased attention towards or away from threat-relevant information will be assessed based on reaction-time based scoring procedures. Higher scores mean greater bias/worse outcomes

SECONDARY OUTCOMES:
Magnitude of respiratory sinus arrhythmia, or variability in heart rate due to respiration rate | Day 1
  Respiratory sinus arrhythmia (RSA), calculated using mobile electrocardiogram, will be assessed during the Trier Social Stress Task, a standardized behavioral assessment of stress. Higher scores mean greater contribution of respiratory rate to heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Dennis, PhD, Principal Investigator — Hunter College, CUNY
Locations (1):
- Hunter College of the City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No